CLINICAL TRIAL: NCT04220385
Title: Comparison Between the Effectiveness of Wii Fit Plus and Core Exercise Program in Improving Core Stability in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tabish Husain Siddiqui, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DUHS/SC/2019/08
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Core Stability
Keywords: Virtual reality exercise; Exercise Therapy/methods; Health Promotion Physical Endurance/physiology; Core Stability
MeSH Terms: interventions — Core Stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wii fit Plus (Active Comparator): This study group will perform the following Wii fit plus exercises
  * Single-Leg Extension
  * Arm and Leg Lift
  * Balance Bridge
  * Single-Leg Twist
  * Single-Leg Reach
  * Sideways Leg Lift
  * Single Arm Stand
  * Torso Twists
  * Plank
  Interventions: Other: Group A
- Core Stability (Active Comparator): This study group will perform the following exercises.
  * Curl-up
  * Side Bridge
  * Bird Dog
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Subjects will perform following exercises, Single Leg Extension, Arm and Leg Lift, Balance Bridge, Single-Leg Twist, Single Leg Reach, Sideways Leg Lift, Single Arm Stand, Torso Twists and Plank exercise with minimum one set and maximum two sets. 30 seconds will be rest time between each set. Subjects will be encouraged to increase the number of repetitions after every 2 weeks, except in Plank exercise in which holding position time will be initially 30 seconds in each set and will be encouraged to increase holding time after every 2 weeks.
  Other Names: Wii fit Plus
  Arms: Wii fit Plus
Other: Group B — Subjects will perform Side Bridge, Bird Dog and Beginner Curl-up exercise in the first three weeks and Side Bridge, Bird Dog and Intermediate Curl-up exercise in the last three weeks. Repetitions per set will be 5, 4, 3 in first two weeks, 7, 6, 5 in third and fourth weeks and 9, 8, 7 in last two weeks. 8-10 seconds will be holding time in each repetition. 30 seconds will be rest time between each set
  Other Names: Core Stability
  Arms: Core Stability

SUMMARY:
This study will compare the effectiveness of core stability and Wii fit plus exercise in improving core stability. Group A will perform Wii fit plus exercises and group B will perform core stability exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 29 years
* Male and female subjects
* Trunk flexor endurance less than 144 seconds in male and 149 seconds in female subjects
* Trunk extensor endurance less than 146 seconds in male and 189 seconds in female subjects
* Flexibility less than 24 cm in male and 27 cm in female.

Exclusion Criteria:

* Weight more than or equal to 150 kg because it is the maximum limit for balance board
* Spinal surgery history,
* Current low back pain
* Performing exercise in routine
* Acute or chronic cardiovascular disease
* Acute or chronic musculoskeletal disease
* Acute or chronic neurological disease.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-11-21 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Change in trunk flexor endurance test | Base line and 6 weeks
  It is expressed in seconds, subject will sit on the test bench and place the upper body against a support with an angle of 60 ° from the test bed. Both the knees and hips will be flexed to 90 °.The arms will be folded across the chest with the hands placed on the opposite shoulder and toes will be placed under toe straps. Subjects will be instructed to maintain the body position while the supporting wedge will be pulled back 10 cm to begin the test. The test will end when the upper body fell below the 60 ° angle.
Change in trunk extensor endurance test | Base line and 6 weeks
  It is recorded in seconds. Subjects will laid prone with the lower body fixed to the test bed at the ankles, knees, and hips and the upper body extended in a cantelevered fashion over the edge of the test bench. The test bench surface will be approximately 25 cm above the surface of the floor. Subjects will rest their upper bodies on the floor before the exertion. At the beginning of the exertion the upper limbs will be held across the chest with the hands resting on the opposite shoulders, and the upper body will be lifted off the floor until the upper torso will be horizontal to the floor. Subjects will be instructed to maintain the horizontal position as long as possible.
Change in sit and reach test | Base line and 6 weeks
  It is expressed in cm.The subject sits without shoes and the soles of the feet flat against a sit-and reach box with the zero mark at the 26 cm. Inner edges of the soles should be 15.2 cm apart.. The subject should slowly reach forward with both hands as far as possible, holding this position approximately 2 s.

CONTACTS AND LOCATIONS:
Overall Officials: Tabish Husain Siddiqui, DPT, MSAPT*, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akuthota V, Ferreiro A, Moore T, Fredericson M. Core stability exercise principles. Curr Sports Med Rep. 2008 Feb;7(1):39-44. doi: 10.1097/01.CSMR.0000308663.13278.69. PMID 18296944
- [Background] Willson JD, Dougherty CP, Ireland ML, Davis IM. Core stability and its relationship to lower extremity function and injury. J Am Acad Orthop Surg. 2005 Sep;13(5):316-25. doi: 10.5435/00124635-200509000-00005. PMID 16148357
- [Background] Reiman MP, Krier AD, Nelson JA, Rogers MA, Stuke ZO, Smith BS. Comparison of different trunk endurance testing methods in college-aged individuals. Int J Sports Phys Ther. 2012 Oct;7(5):533-9. PMID 23091786
- [Background] Sihawong R, Janwantanakul P, Jiamjarasrangsi W. A prospective, cluster-randomized controlled trial of exercise program to prevent low back pain in office workers. Eur Spine J. 2014 Apr;23(4):786-93. doi: 10.1007/s00586-014-3212-3. Epub 2014 Feb 4. PMID 24492949
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] Lopez-Minarro PA, Andujar PS, Rodrnguez-Garcna PL. A comparison of the sit-and-reach test and the back-saver sit-and-reach test in university students. J Sports Sci Med. 2009 Mar 1;8(1):116-22. eCollection 2009. PMID 24150564
- [Background] Zadro JR, Shirley D, Simic M, Mousavi SJ, Ceprnja D, Maka K, Sung J, Ferreira P. Video-Game-Based Exercises for Older People With Chronic Low Back Pain: A Randomized Controlledtable Trial (GAMEBACK). Phys Ther. 2019 Jan 1;99(1):14-27. doi: 10.1093/ptj/pzy112. PMID 30247715
- [Background] Bakar Y, Tugral A, Ozel A, Altuntas YD. Comparison of a 12-Week Whole-Body Exergaming Program on Young Adults: Differentiation in Flexibility, Muscle Strength, Reaction Time, and Walking Speed Between Sexes. Clin Nurs Res. 2020 Sep;29(7):424-432. doi: 10.1177/1054773818797881. Epub 2018 Sep 6. PMID 30188176
- [Background] Neumann S, Meidert U, Barbera-Guillem R, Poveda-Puente R, Becker H. Effects of an Exergame Software for Older Adults on Fitness, Activities of Daily Living Performance, and Quality of Life. Games Health J. 2018 Oct;7(5):341-346. doi: 10.1089/g4h.2017.0079. PMID 30325234
- [Background] Sato K, Kuroki K, Saiki S, Nagatomi R. Improving Walking, Muscle Strength, and Balance in the Elderly with an Exergame Using Kinect: A Randomized Controlled Trial. Games Health J. 2015 Jun;4(3):161-7. doi: 10.1089/g4h.2014.0057. Epub 2015 Jan 28. PMID 26182059
- [Background] Lee D, Lee S, Park J. Effects of indoor horseback riding and virtual reality exercises on the dynamic balance ability of normal healthy adults. J Phys Ther Sci. 2014 Dec;26(12):1903-5. doi: 10.1589/jpts.26.1903. Epub 2014 Dec 25. PMID 25540494
- [Background] Siriphorn A, Chamonchant D. Wii balance board exercise improves balance and lower limb muscle strength of overweight young adults. J Phys Ther Sci. 2015 Jan;27(1):41-6. doi: 10.1589/jpts.27.41. Epub 2015 Jan 9. PMID 25642034
- [Background] Nitz JC, Kuys S, Isles R, Fu S. Is the Wii Fit a new-generation tool for improving balance, health and well-being? A pilot study. Climacteric. 2010 Oct;13(5):487-91. doi: 10.3109/13697130903395193. PMID 19905991
- [Background] Schilling JF, Murphy JC, Bonney JR, Thich JL. Effect of core strength and endurance training on performance in college students: randomized pilot study. J Bodyw Mov Ther. 2013 Jul;17(3):278-90. doi: 10.1016/j.jbmt.2012.08.008. Epub 2012 Sep 15. PMID 23768270